CLINICAL TRIAL: NCT07053215
Title: Efficacy of Argon-Helium Cryoablation Combined With PD-1 Inhibitors in Non-Small Cell Lung Cancer: A Randomized Controlled Trial
Brief Title: Efficacy of Argon-Helium Cryoablation Plus PD-1 Inhibitors in NSCLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Na Li, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZ2023116
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Argon-helium cryoablation; PD-1 inhibitor; Non-small cell lung cancer; Randomized controlled trial; Efficacy; Immune function
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Argon-Helium Cryoablation + PD-1 Inhibitor (Experimental): Patients received argon-helium cryoablation followed by PD-1 inhibitor (Camrelizumab 200 mg IV every 3 weeks for 4 cycles).
  Interventions: Device: Argon-Helium Cryoablation; Drug: Camrelizumab
- PD-1 Inhibitor + Chemotherapy (Active Comparator): Patients received PD-1 inhibitor (Camrelizumab 200 mg IV every 3 weeks) combined with standard platinum-based doublet chemotherapy for 4 cycles.
  Interventions: Drug: Camrelizumab; Drug: Platinum-based doublet chemotherapy

INTERVENTIONS:
Device: Argon-Helium Cryoablation — Procedure performed within 7 days before the first dose of PD-1 inhibitor. CT-guided insertion of cryoprobes into the target tumor. Two freeze-thaw cycles: rapid freeze to -135°C to -145°C for 15-20 minutes, followed by thawing.
  Arms: Argon-Helium Cryoablation + PD-1 Inhibitor
Drug: Camrelizumab — 200 mg intravenously every 3 weeks for 4 cycles.
Drug: Platinum-based doublet chemotherapy — * Non-squamous NSCLC: Pemetrexed (500 mg/m² IV on day 1) plus Carboplatin (AUC 5 mg/mL•min IV on day 1) of each 3-week cycle.
  * Squamous NSCLC: Gemcitabine (1250 mg/m² IV on days 1 and 8) plus Carboplatin (AUC 5 mg/mL•min IV on day 1) of each 3-week cycle.
  * Administered for 4 cycles.
  Arms: PD-1 Inhibitor + Chemotherapy

SUMMARY:
This randomized controlled trial investigated the efficacy and safety of argon-helium cryoablation combined with PD-1 inhibitors compared to PD-1 inhibitors plus chemotherapy for treating non-small cell lung cancer (NSCLC). The study aimed to evaluate differences in survival, tumor response, immune function, and adverse events.

DETAILED DESCRIPTION:
This was a single-center, open-label, randomized controlled trial conducted at the First Hospital of Hebei Medical University, China. Sixty patients with advanced non-small cell lung cancer (NSCLC) were enrolled between December 2020 and December 2023. Patients were randomly assigned (1:1) to either a study group (argon-helium cryoablation combined with PD-1 inhibitor, Camrelizumab) or a control group (PD-1 inhibitor, Camrelizumab, combined with platinum-based doublet chemotherapy). Argon-helium cryoablation was performed prior to PD-1 inhibitor administration in the study group. Both groups received 4 cycles of systemic therapy. The primary endpoints were overall survival (OS) and progression-free survival (PFS). Secondary endpoints included objective response rate (ORR), disease control rate (DCR), changes in immune function markers (CD4+, CD8+, CD4+/CD8+ ratio), and adverse reactions. Patients were followed for up to 1 year. The study aimed to determine if combining cryoablation with PD-1 inhibition offers superior outcomes compared to standard chemo-immunotherapy in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed NSCLC, stage IIIB, IIIC, or IV (AJCC 8th Edition);
* At least one measurable tumor lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1);
* Estimated survival time ≥6 months;
* Receiving argon-helium cryoablation combined with PD-1 inhibitor for the first time at our institution (for study group) or standard chemo-immunotherapy (for control group);
* Unable or unwilling to undergo surgical resection for various reasons;
* Karnofsky Performance Status (KPS) score ≥60;
* Conscious and capable of effective communication;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.

Exclusion Criteria:

* Presence of other active malignant tumors;
* Significant uncontrolled hepatic (total bilirubin >1.5 × upper limit of normal [ULN], AST/ALT >2.5 × ULN or >5 × ULN if liver metastases present) or renal dysfunction (creatinine clearance <50 mL/min);
* Non-primary NSCLC (i.e., metastatic from another site);
* Known allergy or contraindication to study drugs or inability to comply with the treatment plan;
* Coexisting active tuberculosis, uncontrolled systemic infections, or other significant pulmonary diseases that would interfere with treatment or outcome assessment;
* Pregnancy or lactation;
* Severe psychiatric disorders;
* Uncorrected coagulation disorders (e.g., INR >1.5 or platelet count <75 × 109/L);
* Known immunodeficiency syndromes (e.g., HIV infection);
* Symptomatic hemorrhagic pleural effusion requiring urgent intervention;
* Patients who withdrew consent before randomization or were deemed non-compliant by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization until death, assessed through study completion, an average of 1 year.
  Time from randomization to death from any cause.
Progression-Free Survival (PFS) | From randomization until disease progression or death, assessed through study completion, an average of 1 year.
  Time from randomization to disease progression (RECIST 1.1) or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Assessed after 4 cycles of treatment (each cycle is 21 days), at approximately 12 weeks from randomization.
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR) according to mRECIST criteria.
Disease Control Rate (DCR) | Assessed after 4 cycles of treatment (each cycle is 21 days), at approximately 12 weeks from randomization.
  Proportion of patients achieving CR, PR, or Stable Disease (SD) according to mRECIST criteria.
Change in CD4+ T lymphocyte counts | Baseline (Day 1, prior to treatment) and at the end of Cycle 4 (each cycle is 21 days).
  Change in peripheral blood CD4+ T lymphocyte subset counts from baseline.
Change in CD8+ T lymphocyte counts | Baseline (Day 1, prior to treatment) and at the end of Cycle 4 (each cycle is 21 days).
  Change in peripheral blood CD8+ T lymphocyte subset counts from baseline.
Change in CD4+/CD8+ T lymphocyte ratio | Baseline (Day 1, prior to treatment) and at the end of Cycle 4 (each cycle is 21 days).
  Change in the ratio of peripheral blood CD4+ to CD8+ T lymphocytes from baseline.
Incidence and severity of Adverse Events (AEs) | From the first dose of study treatment until 30 days after the last dose of study medication (up to approximately 16 weeks).
  Number and grade of AEs according to NCI-CTCAE v5.0.
1-year Progression-Free Survival Rate | At 1 year from randomization.
  Proportion of patients alive and without disease progression at 1 year from randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China